CLINICAL TRIAL: NCT06652243
Title: An Early Clinical Study to Evaluate the Safety and Efficacy of SN301A Cell Injection in the Treatment of Subjects with Glypican-3 (GPC3)-Positive Advanced Hepatocellular Carcinoma
Brief Title: Clinical Study of SN301A Injection in the Treatment of Hepatocellular Carcinoma
Acronym: SN301A
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Celest Therapeutics Co. Ltd (Unknown); Senti Biosciences (Industry)
Responsible Party: Principal Investigator, Qi Li, Head of Oncology, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SN301A-001
Record Dates: First submitted 2024-10-17; First posted 2024-10-22 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: hepatocellular carcinoma; CAR NK; GPC3
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SN301A CAR NK cell therapy (Experimental): Using the modified "3 + 3" design principle, a total of 3 dose groups are planned,.There were 1 case in the first group and 3 to 6 cases in each of the last two groups ： Dose level 1 (Initial safe dose): 0.5e9 CAR+ NK cells, Dose level 2 (Target effective dose): 1e9 CAR+ NK cells, Dose level 3（Maximum dose）: 2e9 CAR+ NK cells Which are administered once on Days 0, 7, and 14 of each 28 day cycle.
  Interventions: Biological: SN301A

INTERVENTIONS:
Biological: SN301A — SN301A is an investigational off-the-shelf CAR NK cell therapy, armed with calibrated release (cr)IL15, designed to selectively target and treat GPC3 expressing advanced hepatocellular carcinoma.
  Subjects will receive lymphodepletion pretreatment (Fludarabine/Cyclophosphamide), three SN301A intravenous infusions in a cycle (D0, D7, D14), with each subject receiving a maximum of 3 cycles.
  Other Names: Fludarabine; Cyclophosphamide

SUMMARY:
This is a single-arm, open-label study of safety, tolerability, and anti-cancer activity of SN301A (an off-the-shelf CAR NK cell therapy) in patients with glypican-3 (GPC3)-positive advanced hepatocellular carcinoma.

DETAILED DESCRIPTION:
This study is a single-arm, open-label, modified 3+3 dose-escalation early exploratory clinical study to evaluate the safety, tolerability, Pharmacokinetic (PK), and Pharmacodynamic (PD) of SN301A cell injection in the treatment of subjects with glypican-3 (GPC3)-positive advanced hepatocellular carcinoma, and evaluate the efficacy of SN301A cell injection in the treatment of subjects with GPC3-positive advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent (ICF) and capable of complying with protocol-specified visits and related procedures;
2. Age ≥ 18 years and ≤ 70 years, male or female;
3. According to the Guidelines for the Diagnosis and Treatment of Primary Liver Cancer of CSCO in 2024, hepatocellular carcinoma was Diagnosed and GPC3 expression was positive by immunohistochemistry (GPC3 positive was defined as staining positive i.e. ≥ 2 + as defined by Kaseb et al);
4. Barcelona Clinic Liver Cancer (BCLC) stage determined to be unresectable Stage B or C hepatocellular carcinoma, including: disease progression following surgical/local therapy or unsuitable for surgical/local therapy, recurrent or metastatic HCC;
5. Failed at least one prior line of systemic therapy and had used PD-1/L1 and /or TKIs;
6. Child-Pugh A or B 7 points and no history of hepatic encephalopathy;
7. ECOG score 0-1;
8. Life expectancy of no less than 12 weeks;
9. Subjects with at least 1 measurable lesion according to RECIST v1.1 and mRECIST (a lesion that has undergone local therapy such as radiation therapy or interventional therapy cannot be considered measurable unless imaging evidence confirms unequivocal progression of the lesion), RECIST v1.1 i.e., non-nodal lesions ≥ 10 mm in longest diameter and/or nodal lesions ≥ 15 mm in short diameter on CT or MRI; mRECIST refers to non-lymph node measurable disease criteria meeting RECIST v1.1 criteria (hilar lymph nodes must have short axis ≥ 20 mm) and demonstrating intratumoral arterial enhancement on contrast-enhanced CT or MRI ;
10. Subjects must provide either fresh tumor tissue samples that meet the requirements or archival tissue within 2 year prior to signing the ICF;
11. Subject has adequate organ and bone marrow function and meets the following laboratory criteria:

    * Bone marrow function: absolute neutrophil count (ANC) ≥ 1.5e9/L; platelets (PLT) ≥ 75e9/L (transfusion or use of hematopoietic stimulating factors was not acceptable within 14 days prior to Screening);
    * Hemoglobin ≥ 90g/L;
    * Liver function: total bilirubin ≤ 2.5 × ULN; alanine aminotransferase ≤ 5 × ULN; aspartate aminotransferase ≤ 5 × ULN;
    * Renal function: serum creatinine ≤ 1.5 × ULN, or creatinine clearance ≥ 60 mL/min (calculated using the Cockcroft-Gault formula);
    * Coagulation: International normalized ratio (INR) ≤ 1.5 × ULN, activated partial thromboplastin time (APTT) ≤ 1.5 × ULN (INR between 2.0 and 3.0 is required for subjects receiving prophylactic anticoagulant therapy);
12. Men and women of childbearing potential must agree to use effective contraception from signing the ICF until one year after the last cell infusion and must have a negative serum pregnancy test at screening for women of childbearing potential.

Exclusion Criteria:

1. Metastases to central nervous system, including brain metastases and/or meningeal metastases;
2. Prior bone marrow or organ transplant (including but not limited to liver transplant) or waiting for transplant;
3. Previous or concurrent history of other malignancies, except for carcinoma in situ of the uterine cervix that has been cured and has not recurred for at least 2 years before screening, noninvasive basal cell or squamous cell skin cancer, or ductal carcinoma in situ after radical treatment for localized prostate cancer and radical resection;
4. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and HBV DNA > 500 IU/mL (lower limit of detection; HBV DNA ≤ 500 IU/mL, lymphodepletion pretreatment requires antiviral therapy for at least 14 days before treatment and can be enrolled if antiviral therapy is continued during the study); hepatitis C virus (HCV) antibody positive and HCV RNA positive; human immunodeficiency virus (HIV) antibody positive; syphilis antibody positive;
5. HLA antibody positive subjects, including weak positive, positive and strong positive (except those with HLA typing different from SN301A cell injection products);
6. Prior treatment with other cellular products or GPC3-targeted agents;
7. Received any fluoropyrimidine chemotherapeutic agents or small-molecule targeted agents within 14 days or 5 half-lives (whichever is shorter) prior to signing the ICF; received any antineoplastic biological agents or non-fluoropyrimidine chemotherapeutic agents within 28 days prior to signing the ICF; received wide-range radiotherapy within 28 days prior to signing the ICF, received local radiotherapy for non-target lesions to relieve symptoms within 14 days prior to signing the ICF; received traditional Chinese medicine/Chinese herbal medicine and local interventional therapy with anti-tumor indications within 14 days prior to signing the ICF;
8. Adverse events resulting from prior anticancer therapy have not recovered to Grade 1 or baseline, except for alopecia, Grade 2 peripheral neurotoxicity, hypothyroidism stabilized by hormone replacement;
9. Subjects who have received attenuated live vaccine immunization within 28 days prior to signing ICF or need to receive attenuated live vaccine immunization during the study;
10. Major surgical treatment (except liver mass biopsy) within 28 days prior to signing the ICF, or the need for major surgical treatment during the study;
11. Requiring chronic systemic corticosteroids (at doses ≥ 10 mg/day prednisone or equivalent) or other immunosuppressive medications within 14 days prior to the first study drug infusion or during the study, except for inhaled or topical use;
12. Subjects with fungal, bacterial, viral, tuberculosis or other infection requiring systemic anti-infective treatment within 14 days prior to signing the ICF;
13. Patients with active or previous autoimmune diseases that may recur, such as systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vasculitis, psoriasis, etc.;
14. Previous or current interstitial lung disease, pneumonoultra microscopic pneumonitis, radiation pneumonitis, severely impaired pulmonary function, etc.;
15. Third space effusion that is not clinically well controlled before screening, such as pleural effusion and ascites that cannot be controlled by drainage or other methods;
16. History of serious cardiovascular and cerebrovascular diseases, including but not limited to in:

    * Patients with severe heart rhythm or conduction abnormalities, such as ventricular arrhythmia requiring clinical intervention, grade II-III atrioventricular block;
    * QT interval corrected by Fridericias formula (QTcF) prolongation > 450 ms for males; > 470 ms for females;
    * Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other ≥ Grade 3 cardiovascular or cerebrovascular event within 6 months prior to Screening;
    * Presence of heart failure of New York Heart Association (NYHA) Functional Class ≥ II or left ventricular ejection fraction (LVEF) > 50%;
    * Clinically uncontrolled hypertension, systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg.
17. Patients with history of pulmonary embolism or severe lower extremity deep venous thrombosis requiring interventional treatment such as inferior vena cava filter implantation or therapeutic dose of anticoagulants at screening;
18. Investigator assessment of intrahepatic tumor mass greater than 50% of the entire liver, or tumor thrombus invading major vessels such as the main portal vein, superior mesenteric vein, or inferior vena cava causing complications such as portal hypertension or associated clinical risks;
19. Subject is participating in another interventional clinical study;
20. Pregnant or lactating women;
21. Subjects with other conditions that, in the opinion of the investigator, could affect compliance or unsuitability for participation in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities | 28 days post SN301A infusion.
  Incidence of DLT after the first infusion of SN301A cell injection
Incidence and severity of adverse events (AEs)and serious adverse events (SAEs) (Safety and Tolerability) | Through study completion, up to 2 years
  Any untoward medical event that occurs after a subject has administered an investigational product, which may be manifested as a symptom, sign, disease or laboratory abnormality but does not necessarily have a causal relationship with the investigational product.

SECONDARY OUTCOMES:
Objective response rate (ORR) after SN301A infusion | Through study completion, up to 2 years
  Efficacy results of SN301A
Disease control rate (DCR) after SN301A infusion | Through study completion, up to 2 years
  Efficacy results of SN301A
Duration of response (DOR) after SN301A infusion | Through study completion, up to 2 years
  Efficacy results of SN301A
Progression-free survival (PFS) after SN301A infusion | Through study completion, up to 2 years
  Efficacy results of SN301A
Overall survival (OS) after SN301A infusion | Through study completion, up to 2 years
  Efficacy results of SN301A
Concentration of alpha fetoprotein (AFP) after SN301A infusion | Through study completion, up to 2 years
  Efficacy results of SN301A
Concentration of abnormal prothrombin after SN301A infusion | Through study completion, up to 2 years
  Efficacy results of SN301A
Concentration of carbohydrate antigen 19-9 after SN301A infusion | Through study completion, up to 2 years
  Efficacy results of SN301A
PK parameters of CAR NK cells in peak peripheral blood (Cmax) after SN301A infusion | Through study completion, up to 2 years
  Pharmacokinetic (PK) results of SN301A
PK parameters of CAR NK cells in time to peak peripheral blood (Tmax) after SN301A infusion | Through study completion, up to 2 years
  Pharmacokinetic (PK) results of SN301A
PK parameters of CAR NK cells in half-life (t 1/2) after SN301A infusion | Through study completion, up to 2 years
  Pharmacokinetic (PK) results of SN301A
PK parameters of CAR NK cells in area under the concentration versus time curve (AUC) after SN301A infusion | Through study completion, up to 2 years
  Pharmacokinetic (PK) results of SN301A
Levels of cytokines (IL-6, IFN-γ, TNF-α, IL-15) in peripheral blood after SN301A infusion | Through study completion, up to 2 years
  Pharmacokinetic (PK) results of SN301A

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No